CLINICAL TRIAL: NCT01984710
Title: Deep Brain Stimulation for Treatment Resistant Depression: Exploration of Local Field Potentials (LFP) With the Medtronic Activa Primary Cell + Sensing (PC+S) "Brain Radio" System
Brief Title: Deep Brain Stimulation for Treatment Resistant Depression With the Medtronic Activa PC+S
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Hope for Depression Research Foundation (Other); The Dana Foundation (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Patricio Riva Posse, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00066843; 5UH3NS103550 (NIH)
Record Dates: First submitted 2013-09-23; First posted 2013-11-15 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Treatment Resistant Depression
Keywords: Treatment Resistant Depression; Deep Brain Stimulation; Psychiatry; Neuro Surgery
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- DBS for Treatment Resistant Depression (Experimental): DBS for TRD: Exploration of LFP with the Medtronic Activa PC+S "Brain Radio" system
  Interventions: Device: Medtronic Activa PC+S System

INTERVENTIONS:
Device: Medtronic Activa PC+S System
  Other Names: Medtronic Inc

SUMMARY:
The goal of this study is to use the Activa Primary Cell + Sensing (PC+S) device to study Latent Field Potential (LFP) in the brains of people with Treatment Resistant Depression (TRD) before and during active stimulation. The ultimate goal is to understand the neural network that causes TRD and the changes that DBS cause in that network that results in the antidepressant effects.

DETAILED DESCRIPTION:
Major depressive disorder is a common disease. For many people, conventional treatments such as antidepressants are very helpful in relieving the symptoms of this condition. But as many as 30% of patients with depression have less than a full response or become resistant to conventional treatments. When treatment resistance develops, the depression becomes a chronic disease with a very significant burden of morbidity and mortality. The reasons that some patients develop Treatment Resistant Depression (TRD) are not known. One current theory for depression is that it results from the dysfunction of a network of regions in the brain and that in treatment resistant patients the network is permanently stuck in the dysfunctional state. We have been investigating an experimental treatment for treatment resistant depression (TRD), based on this network theory known as subcallosal deep brain stimulation (SCC DBS). This treatment involves placement of electrodes in a specific region of the brain (subcallosal cingulate cortex, area 25) and then stimulating that area with electricity, which resets the regulation of the network resulting in a significant antidepressant response. While still experimental our results suggest this may eventually be a useful treatment for some patients with TRD. The experiment described in this application is to use a new DBS device that can record the electrical activity in the brain around the site of stimulation. The electrical activity is known as Latent Field Potential (LFP) and is a reflection of the activity if the neural network. The new DBS device is an experimental device that has not been approved by the Food and Drug Administration (FDA), but allows for simultaneous recording of LFP while stimulation is being delivered. The device is manufactured by Medtronics and is known as Activa Primary Cell + Sensing(PC+S), but because it can be used to record the brain electrical activity it is also known as "the Brain Radio". The Brain Radio is based on an approved device commonly used for DBS for other conditions that has the added sensor capacity. The stimulation system is identical to that in the approved device. The goal of this investigation is to use the Brain Radio to study LFP in the brains of people with TRD before and during active stimulation. The ultimate goal is to understand the neural network that causes TRD and the changes that DBS cause in that network that results in the antidepressant effects. We will recruit 10 patients with advanced TRD and implant them with the Brain Radio system. The recording system will be to record LFP over 3 years, while patients receive stimulation. A brief discontinuation study will be conducted after 6 months of stimulation when the device will be turned off and patterns of LFP changes will be recorded. All LFP measures will be correlated with the primary clinical response outcome metric, the Hamilton Depression Rating Scale. The knowledge gained with this experiment will be invaluable to understanding the basic pathology of depression and the antidepressant response. This is a unique, first in humans test of this device and as such the results are expected to impact our understanding of depression at a fundamental basis.

Deep brain stimulation of the subcallosal cingulate white matter (SCC25 DBS) has been investigated as a new interventional strategy for treatment resistant depression (TRD). In addition to growing evidence of long-term antidepressant efficacy with chronic stimulation, immediate changes in mood, attention, and psychomotor speed during intra-operative testing have been repeatedly observed. These acute, electrode contact-specific behavioral effects have successfully guided selection of the optimal contact for chronic DBS. The presence of intraoperative behavioral effects is often predictive of long-term outcome. It is clear that sustained high frequency stimulation appears to be required to maintain the antidepressant response long-term, as discontinuation even after several years of remission is associated with deterioration and return of depression symptoms over several weeks. Imaging studies examining effects of chronic SCC25 DBS using positron emission tomography (PET) demonstrate changes in blood flow and metabolism both in the vicinity of the DBS target, and remotely in frontal cortex, ventral striatum, hypothalamus and amygdala/hippocampus. These findings, combined with more recent diffusion tensor imaging (DTI) studies, provide evidence of the anatomical and functional extent of regional changes mediating antidepressant effects of DBS over time [5-6].

Brain changes mediating the observed intra-operative behavioral changes or discontinuation-precipitated relapse are unknown. To date, none of the studies have been able to address explicit mechanisms of DBS for TRD at the neuronal level, during chronic stimulation. It is possible to make measurements of neuronal activity with available recording systems only during intraoperative testing. Given that TRD requires chronic stimulation to achieve full remission, characterization of changes in neural activity throughout the duration of stimulation and development of therapeutic response will be invaluable in further developing and refining this treatment modality. Furthermore, tracking of neural changes and their behavioral correlates with chronic stimulation and controlled discontinuation would allow characterization of physiologic markers for potential use as feedback signals for further treatment development and optimization.

This set of new experiments will build on past experience of utilizing SCC25 DBS in patients with TRD to explore potential neural correlates of antidepressant response. This will be done using the ActivaPC+S, which is a prototype DBS system developed by Medtronic that combines conventional DBS brain electrodes and pulse generator with a sensing device that can chronically read, record and download the electrical brain activity known as Local Field Potential (LFP) at the brain area surrounding the DBS electrode. These recordings can be downloaded from the implanted device with an external antenna device similar to the device used to control the pulse generator. Given the ability to record LFP locally in the brain and to transmit this information to a receiving station the ActivaPC+S device is referred to as the "Brain Radio".

The ActivaPC+S, "Brain Radio" device is an experimental system currently not approved by the FDA. This device is based on the ActivaPC system, which has FDA approval for use in Parkinson's disease, Essential Tremor and has Humanitarian Device Exemption (HDE) for Dystonia. The ActivaPC also has an HDE for use in intractable Obsessive Compulsive Disorder (OCD). The Brain Radio has sensing technology in addition to the standard stimulation capacity of the approved device that allows for real time recording of LFP in the anatomical location of the electrode both during active stimulation and when stimulation is off. As such this is a very powerful research tool that will facilitate investigation of the neuronal changes associated with antidepressant response to chronic DBS. This will be the first ever use of this unique, cutting edge system in human patients with treatment resistant depression and has the potential to provide unprecedented insight into the fundamental neuronal processes that underlie depressive illness and antidepressant response.

Hypothesis 1: Aberrant oscillations in the SCC-prefrontal circuitry are present in TRD patients. SCC25 DBS exerts its therapeutic effects by altering these network dynamics. Behavioral improvements in TRD patients treated with SCC25 DBS will correlate with discernible LFP changes at specific DBS electrode contacts, both acutely and chronically.

Hypothesis 2: Stable maintenance of stimulation-induced LFP changes is required for sustained antidepressant response, with loss of these changes heralding impending depression relapse.

This study will test these hypotheses in 10 TRD patients via recording LFPs with the ActivaPC+S system throughout the course of chronic SCC25 DBS. Measures of SCC LFP oscillatory activity will be correlated with clinical measures of antidepressant response and with scalp EEG signals.

OBJECTIVES Experiment #1: To quantify electrophysiological changes, behavioral correlates and EEG changes in the month following implantation when the stimulator is turned OFF.

Experiment #1A: To characterize the LFP changes for 48 hours post op in response to the brief, acute stimulation the patient receives during the implantation procedure Experiment #1B: To characterize the changes in LFP patterns in the month after implantation and to establish a baseline before chronic stimulation is initiated. The Activa PC+S system will be utilized to record LFP during this phase of the protocol.

Experiment #2: The stimulator will be turned on 1 month after implantation. This experiment will occur on the day of stimulation initiation. Clinical data will be recorded and LFP changes will be captured by the Activa PC+S system and scalp EEG. The stimulator will be cycled through a series of different frequency and current settings while LFPs are recorded.

Experiments #3: To quantify LFP changes in response to chronic high frequency SCC25 stimulation and to correlate change patterns with long-term antidepressant response and EEG patterns. Stimulation will be initiated one month after implantation and maintained chronically for the subsequent 6 months. Clinical assessments, LFP and scalp EEG will be routinely recorded during this 6-month period.

Experiment #4: To quantify LFP changes when the stimulation is briefly stopped (1 week) after 6 months of chronic stimulation. Correlation will be made between LFP, clinical/ symptomatic changes and EEG patterns.

Experiment #5: To quantify LFP changes over the extended period of exposure to chronic high frequency SCC25 stimulation. Clinical response and EEG patterns will be recorded every 6 months and compared to LFP over the battery life of the ActivaPC+S system; currently estimated at 3 to 5 years after initiation of stimulation.

The primary clinical outcome metric is the Hamilton Depression Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent.
* Agrees to relocate to the Atlanta Metro region for the duration of the acute phase of the investigation (approximately 8-10 months) and to return regularly for clinical and research assessments
* Current Major Depressive Episode (MDE), either Major Depressive Disorder single episode or recurrent type
* Current depressive episode of at least two years duration or a history of more than 4 lifetime depressive episodes
* Minimum score at study entry of 20 on the 17-item Hamilton Depression Rating Scale (HDRS-17)
* Average pre-operative HDRS-17 score of 20 or greater (averaged over four weekly pre-surgical evaluations during the four weeks prior to surgery) and an average pre-operative HDRS-17 score no more than 30% lower than the baseline screening HDRS-17 score
* A maximum Global Assessment of Functioning of 50 or less
* Failure to respond to a minimum of four different antidepressant treatments, including at least three medications from at least three different drug classes, evidence-based psychotherapy or electroconvulsive therapy (ECT) administered at adequate doses and duration during the current episode
* Failure or intolerance of an adequate course of electroconvulsive therapy (ECT) during any episode
* On stable antidepressant medication
* Have an established outpatient psychiatrist and be willing to sign a written release to allow study investigators to give and receive information from this psychiatrist

Exclusion Criteria:

* Inability/ refusal to sign written informed consent
* Refusal or inability to relocate to Atlanta Metro region for acute phase of protocol or to return for regular assessments in long term follow up
* Inability to tolerate general anesthesia
* Significant cerebrovascular risk factors or a previous stroke, documented major head trauma or neurological disorder
* Other currently active clinically significant Axis I psychiatric diagnosis including bipolar disorder, schizophrenia, panic disorder, obsessive-compulsive disorder, generalized anxiety disorder or post-traumatic stress disorder
* Current psychotic symptoms
* Evidence of global cognitive impairment
* Substance abuse or dependence not in full, sustained remission
* Active suicidal ideation with intent; suicide attempt within the last six months; more than three suicide attempts within the last two years
* Pregnancy or plan to become pregnant during the study period
* General contraindications for DBS surgery (cardiac pacemaker/defibrillator or other implanted devices)
* Inability or unwillingness to comply with long-term follow-up
* History of intolerance to neural stimulation of any area of the body
* Participation in another drug, device or biologics trial within the preceding 30 days prior to initial screening
* Conditions requiring repeated MRI scans
* Conditions requiring diathermy
* Conditions requiring anticoagulant medication
* Terminal illness associated with expected survival of <12 months

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Activa PC+S Local Field Potential (LFP) Recordings | From Day 1, up to 3 years
  Electrophysiological changes in response to stimulation will be quantified. Continuous Activa PC+S Local Field Potential (LFP) recordings will be monitored from Day 1 post-op until the battery is depleted, which is anticipated to be after approximately 2-3 years.
Change in Hamilton Depression Rating Scale-17 Score | Baseline; Recovery period with stimulation off: 24 hours post-operative, Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The Hamilton Depression Rating Scale (HDRS-17) contains 17 items that are scored from 0 to 2, 3, or 4, where 0 is lack of difficulty and the highest number for an item is the most extreme difficulty. Total scores can range from 0 to 52 where higher scores represent greater symptom severity. Scores of 0-7 are considered normal, scores of 8-16 indicates mild depression, scores of 17-23 indicate moderate depression, and scores of 24 and greater indicate severe depression.

SECONDARY OUTCOMES:
Change in Hamilton Anxiety Rating Scale (HAM-A) Score | Baseline; Recovery period with stimulation off: 24 hours post-operative, Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The HAM-A is a 14-item clinician-administered scale that assesses the severity of symptoms of anxiety on a 5-point scale where 0 = not present and 4 = very severe. Total scores range from 0 to 56 with higher scores indicating greater anxiety.
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) Score | Baseline; Recovery period with stimulation off: 24 hours post-operative, Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The MADRS is a 10-item scale where the survey administrator rates the participant on a variety of aspects related to depression (such as apparent sadness, tension, and pessimistic thoughts) based on a clinical interview. Responses are provided on a scale of 0 to 6 where 0 signifies no difficulties in this area and 6 signifies severe difficulty. Total scores range from 0 to 60 with higher scores indicating greater severity of depression.
Change in Beck Depression Inventory (BDI-2) Score | Baseline; Recovery period with stimulation off: 24 hours post-operative, Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The BDI-2 is a self-report measure assessing depressive symptom severity. Total scores ranges from 0 to 63, with a higher score indicating a higher level of depression.
Change in Beck Anxiety Inventory (BAI) Score | Baseline; Recovery period with stimulation off: 24 hours post-operative, Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The BAI is a 21-item self-report measure of anxiety symptoms, rated on a 4-point Likert scale modified to be based on the patient's experience in the past week. Items are rated from 0 = not at all to 3 = severely. Total scores range from 0 to 63 and higher scores indicate greater anxiety.
Change in Inventory of Depressive Symptomatology - Subject Rated (IDS-SR) Score | Baseline; Recovery period with stimulation off: Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The Inventory of Depressive Symptomatology-Self-Report (IDS-SR) is a 30-item questionnaire asking respondents about symptoms of depression that they have experienced in the past 7 days. Each item is scored on a 4-point scale where 0 means that the symptom is absent and 3 means that the symptom is very strongly felt. Total scores can range between 0 and 84 and higher scores indicate more severe symptoms of depression.
Change in Young Mania Rating Scale (YMRS) Score | Baseline; Recovery period with stimulation off: 24 hours post-operative, Week 4; Stimulation phase: as needed up to week 30; Naturalistic follow up: as needed for up to 10 years
  The Young Mania Rating Scale (YMRS) is an11-item instrument assessing manic symptoms in the previous 48 hours. Responses are given on a scale from 0 to 4 or 0 to 8, where 0 = the symptom is absent or at a normal level and the highest score (4 or 8) = the symptom is extreme. Total scores range from 0 to 60 where higher values indicate increased symptoms of mania.
Change in Patient Global Impression of Severity (PGI-S) Score | Baseline, Recovery period with stimulation off: 24 hours post-operative, Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The Patient Global Impression of Severity (PGI-S) instrument is a single-item assessment of self-rated severity of a specific condition. Responses are given on a 4-point scale where 1 = the condition is normal and 4 = the condition is severe.
Change in Patient Global Impression of Improvement (PGI-I) Score | Recovery period with stimulation off: 24 hours post-operative, Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The Patient Global Impression of Improvement (PGI-I) instrument is a single-item assessment of self-rated improvement of a specific condition. Participants indicate how their condition has changed from baseline on a 7 point scale where 1 = much better, through 7 = very much worse.
Change in Clinical Global Impression for Severity (CGI-S) Score | Baseline; Recovery period with stimulation off: 24 hours post-operative, Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The Clinical Global Impression of Severity (CGI-S) Scale is a clinician's assessment of patient's severity of illness. The score ranges from 1 = normal, not at all ill to 7 = among the most extremely ill patients
Change in Clinical Global Impression - Improvement (CGI-I) | Recovery period with stimulation off: 24 hours post-operative, Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The Clinical Global Impression for Improvement (CGI-I) Scale is a clinician's assessment of a patient's change in condition from baseline.The score ranges from 0 = not assessed, 1 = very much improved, through 7 = very much worse.
Change in Number of Participants with Medication Adjustments | Baseline; Recovery period with stimulation off: Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  Types of medications and doses that participants are taking will be reviewed at study visits.
Change in Positive and Negative Affect Scale (PANAS) Score | Baseline; Recovery period with stimulation off: 24 hours post-operative, Weeks 1, 2, 3, 4; Stimulation phase: every 1-2 weeks up to week 30; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The Positive and Negative Affect Scale (PANAS) consists of 10 positively and 10 negatively valanced word items. Items are rated by the participant for the extent they are feeling this "right now" on a scale of 1- slightly or not at all through 5- extremely. Total scores can range from 10-50, with higher scores representing higher levels of positive effect and lower scores having negative effect.
Change in Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Score | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  Perceived quality of life and general well being was assessed using the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF). The Q-LES-Q-SF is a 16-item questionnaire asking participants to rate how satisfied they have been with heath related qualities on a 5-point scale where 1 = very poor and 5 = very good. Raw scores of the Q-LES-Q-SF range from 14 to 70 and higher scores indicate higher life enjoyment and satisfaction.
Change in Health and Labor Questionnaire (HLQ) Absence from Paid Work Module | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  The HLQ assesses the relationship between illness and treatment and work performance. The HLQ includes four modules examining absences from work, reduced productivity at paid work, unpaid work, and impediments to paid and unpaid labor. The absence from work module asks respondents who work for pay how many days in the past two weeks they missed work due to health problems.
Change in Health and Labor Questionnaire (HLQ) Reduced Productivity at Paid Work Module | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  The HLQ assesses the relationship between illness and treatment and work performance. The HLQ includes four modules examining absences from work, reduced productivity at paid work, unpaid work, and impediments to paid and unpaid labor. The reduced productivity at paid work module examines reduced efficiency when people must go to work with their illness. Respondents who work while ill answer 6 questions rating their productivity on a 4-point scale where 1 = never and 4 = always. Total scores for this section range from 6 to 24 and higher scores indicate greater impacts to productivity.
Change in Health and Labor Questionnaire (HLQ) Unpaid Work Module | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  The HLQ assesses the relationship between illness and treatment and work performance. The HLQ includes four modules examining absences from work, reduced productivity at paid work, unpaid work, and impediments to paid and unpaid labor. Respondents who do not work for pay are asked about the number of hours they spent during the past two weeks doing household work, shopping, odd jobs and chores, and caring for their own children. They are also asked if other people (family, neighbors, or paid help) had to perform those tasks due to the respondent's health problems. The number of hours of unpaid work, normally performed by the participant, that were completed by others due to health problems of the participant are examined.
Change in Health and Labor Questionnaire (HLQ) Impediments to Paid and Unpaid Labor Module | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  The HLQ assesses the relationship between illness and treatment and work performance. The HLQ includes four modules examining absences from work, reduced productivity at paid work, unpaid work, and impediments to paid and unpaid labor. In the impediments to paid and unpaid labor module, respondents are asked if they have performed household work at home, shopping, odd jobs and chores, and doing things for their own children in the past two weeks. Possible responses are "did do, hindered" (scored as 1), "did do, not hindered (scored as 0), "did not do, due to health problems" (scored as 2), and "did not do, due to other reasons" (scored as 0). Total scores range from 0 to 8 where higher scores indicate more impediments to performing paid and unpaid work.
Change in Stressful Life Events (SLE) Questionnaire Score | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  The Stressful Life Events (SLE) Questionnaire is a 46-item instrument assessing 11 domains of Home Life, Financial Problems, Social Relations, Personal Conflicts, Job Conflicts, Educational Concerns, Job Security, Loss and Separation, Sexual Life, Daily Life, and Health Concerns. Respondents self-report the frequency and intensity of life stressors on a 6-point scale where 0 = never and 5 = very severe. Total scores range from 0 to 230 where higher scores indicate greater life stress.
Change in Beck Hopelessness Scale (BHS) Score | Baseline; Recovery period with stimulation off: Weeks 1, 2, 3, 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 1 to 6 months for up to 10 years
  The Beck Hopelessness Scale (BHS) assesses aspects of hopelessness of feelings about the future, loss of motivation, and expectations. The BHS has 20 true/false asking respondents about negative expectations about the future over the previous week. Total scores range from 0 to 20 where higher scores indicate increased hopelessness.
Change in Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  The C-SSRS asks respondents up to 6 questions, depending on the answers to certain questions. Respondents answer "yes" or "no" to questions about thoughts or plans of suicide. Rather than a total score, the survey results indicate if a person is feeling suicidal or not. Any responses of "yes" to the C-SSRS questions are considered a positive response, indicating that the participant is experiencing thoughts of suicide or has exhibited suicidal behaviors.
Change in Zung Self-Rating Depression Scale (SDS) Score | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  During the Self-Rating Depression Scale (SDS) assessment, respondents answer 20 questions about emotions and physical symptoms during the past several days. Responses are given on a 4 point scale where 1 = a little of the time and 4 = most of the time. Total raw scores range from 20 to 80. Total scores can also be converted to an SDS index score which ranges from 25 to 100. Index scores of 25-49 are in the normal range, scores of 50-59 indicate mild depression, scores of 60-69 indicate moderate depression, and scores of 70 and above indicate severe depression.
Change in Global Assessment of Functioning (GAF) Scale Score | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  The Global Assessment of Functioning (GAF) is a scale assessing the severity of mental illness by rating how much symptoms impact daily life. Clinicians score the participant on a scale from 0 to 100 where higher scores indicate increased ability to manage activities of daily life.
Change in Number of Participants Meeting Major Depressive Episode Criteria | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  Categorical definition of presence of major depressive episode (MDE) will be by the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) diagnostic criteria as determined by clinician interview. Depressive relapse will defined as meeting DSM-IV criteria for a MDE (i.e., meeting 5 of 9 DSM-IV criteria for 2 consecutive weeks with at least one symptom being depressed mood or anhedonia) in the absence of a 2-month period of remission. Recurrence will be defined as meeting DSM-IV criteria for a MDE following at least a 2-month period of remission.
Change in 9-item Patient Health Questionnaire (PHQ-9) Score | Baseline; Recovery period with stimulation off: Week 4; Stimulation phase: Weeks 4, 12, 24; Naturalistic follow up: every 6 months for up to 10 years
  Depressive symptoms are assessed by the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a 9-item scale where respondents indicate how much they are bothered by certain problems on a 4-point scale where 0 = not at all and 3 = nearly every day. Total scores range from 0 to 27 with degree of depression considered minimal for scores between 0-4, mild for scores of 5-9, moderate for scores of 10-14, moderate to severe for scores 15-19, and severe for scores of 20-27.

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Riva Posse, MD, Principal Investigator — Emory University; Helen Mayberg, MD, Principal Investigator — Emory University and Mount Sinai; Christopher Rozell, PhD, Principal Investigator — Georgia Institute of Technology
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Alagapan S, Choi KS, Heisig S, Riva-Posse P, Crowell A, Tiruvadi V, Obatusin M, Veerakumar A, Waters AC, Gross RE, Quinn S, Denison L, O'Shaughnessy M, Connor M, Canal G, Cha J, Hershenberg R, Nauvel T, Isbaine F, Afzal MF, Figee M, Kopell BH, Butera R, Mayberg HS, Rozell CJ. Cingulate dynamics track depression recovery with deep brain stimulation. Nature. 2023 Oct;622(7981):130-138. doi: 10.1038/s41586-023-06541-3. Epub 2023 Sep 20. PMID 37730990
- [Derived] Riva-Posse P, Crowell AL, Wright K, Waters AC, Choi K, Garlow SJ, Holtzheimer PE, Gross RE, Mayberg HS. Rapid Antidepressant Effects of Deep Brain Stimulation and Their Relation to Surgical Protocol. Biol Psychiatry. 2020 Oct 15;88(8):e37-e39. doi: 10.1016/j.biopsych.2020.03.017. Epub 2020 May 14. No abstract available. PMID 32418613
- [Derived] Veerakumar A, Tiruvadi V, Howell B, Waters AC, Crowell AL, Voytek B, Riva-Posse P, Denison L, Rajendra JK, Edwards JA, Bijanki KR, Choi KS, Mayberg HS. Field potential 1/f activity in the subcallosal cingulate region as a candidate signal for monitoring deep brain stimulation for treatment-resistant depression. J Neurophysiol. 2019 Sep 1;122(3):1023-1035. doi: 10.1152/jn.00875.2018. Epub 2019 Jul 17. PMID 31314668

DOCUMENTS (1):
  • Informed Consent Form (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT01984710/ICF_000.pdf